CLINICAL TRIAL: NCT02522858
Title: Anticholinergic Premedication for Sedation With Dexmedetomidine During Spinal Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sira Bang (Other)
Responsible Party: Sponsor-Investigator, Sira Bang, Seoul Paik Hospital, Seoul, Korea, Inje University
Organization: Inje University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IIT-2015-101
Record Dates: First submitted 2015-08-05; First posted 2015-08-13 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2016-01

CONDITIONS: Bradycardia
Keywords: premedication; dexmedetomidine; anesthesia, spinal
MeSH Terms: conditions — Bradycardia | interventions — Atropine; Dexmedetomidine; Ephedrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Placebo (Placebo Comparator): After fixation of the block level of spinal anesthesia, and just before starting dexmedetomidine, normal saline 0.5mL would be injected intravenously.
  Interventions: Drug: Dexmedetomidine; Drug: Ephedrine
- Atropine (Experimental): After fixation of the block level of spinal anesthesia, and just before starting dexmedetomidine, ,atropine 0.03mg/kg would be injected intravenously.
  Interventions: Drug: Atropine; Drug: Dexmedetomidine; Drug: Ephedrine

INTERVENTIONS:
Drug: Atropine — To evaluate the effectiveness of atropine on prevention bradycardia,atropine 0.01~0.03mg/kg up to 0.5mg would be injected intravenously just before starting loading dose of dexmedetomidine in group A.
  During operation, heart rate decreasing 30% from initial heart rate or under 40/min would be regarded as bradycardia needing treatment, and atropine 0.5mg will be injected intravenously. This intervention would be applied to both group.
  Arms: Atropine
Drug: Dexmedetomidine — Dexmedetomidine is a highly selective a2 adrenergic receptor antagonist used as sedative agent. After confirming the fixation level of spinal anesthesia, the loading dose(0.6ug/kg) of dexmedetomidine which is diluted with normal saline as 4ug/mL would be started for 10 minutes.Maintenance dose(0.25ug/kg/hr) would be continued after loading dose.
Drug: Ephedrine — Systolic blood pressure decreasing 30% from basal blood pressure or under 90 mm Hg would be regarded as hypotension needing treatment, and ephedrine 5mg will be injected intravenously.

SUMMARY:
Dexmedetomidine is a selective α2 adrenergic receptor antagonist, which has little effect on respiratory suppression used as sedative agent. Also, dexmedetomidine has been reported to prolong the anesthesia time when used with patients undergoing spinal anesthesia. However, dexmedetomidine has sympathetic effect which can cause hypotension and bradycardia dose dependently. Therefore, this study is aimed to evaluate the effectiveness of premedication of anticholinergic agents on vital sign in patients undergoing spinal anesthesia.

DETAILED DESCRIPTION:
Before entering the operation room, patients are randomized in one group (A or C). For sedative premedication, all patients will be injected intramuscularly with midazolam 1mg. After entering the operation room, all patients will be monitored blood pressure, ECG and oxygen saturation. Before induction of spinal anesthesia, all patients will be loaded with plasma solution 5mL/kg. After induction of spinal anesthesia, block level will be checked. After fixation of block level, the loading dose(0.6ug/kg) of dexmedetomidine which is diluted with normal saline as 4ug/mL would be started for 10 minutes. However, just before starting dexmedetomidine,atropine .01~0.03mg/kg up to 0.5mg would be injected in group A. Otherwise normal saline 0.5mL would be injected in group C. The syringed would be blinding not to be noticed. After loading of dexmedetomidine, the diluted solution would be injected with 0.25ug/kg/hr until the end of the surgery. Every patients undergoing sedation would be applied the oxygen by nasal prong.

The heart rate decreasing 30% from initial heart rate or under 40/min would be regarded as bradycardia needing treatment, and atropine 0.5mg will be injected intravenously. Systolic blood pressure decreasing 30% from basal blood pressure or under 90 mm Hg would be regarded as hypotension needing treatment, and ephedrine 5mg will be injected intravenously. The number of medication treated would be noted.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergoing spinal anesthesia with sedation over 19 years old.

Exclusion Criteria:

* Patients who are contraindicated of spinal anesthesia such as hypovolemic status, coagulation disorder, infection of tapping site, pregnancy, heart problem, history of drug allergy, drug abuser, anemia, headache and medication of antipsychotic drugs.
* Patiensts who are contraindicated of atropine such as glaucoma, voiding difficulty due to prostate hyperplasia, heart disease, ulcerative colitis, hyperthyroidism and fever.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-08; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
The incidence of bradycardia | 30miniutes from starting dexmedetomidine with loading dose
  The heart rate decreasing 30% from initial heart rate or under 40/min would be regarded as bradycardia needing treatment, and atropine 0.5mg will be injected intravenously.

SECONDARY OUTCOMES:
The incidence of hypotension | 30miniutes from starting dexmedetomidine with loading dose
  Systolic blood pressure decreasing 30% from basal blood pressure or under 90 mm Hg would be regarded as hypotension needing treatment, and ephedrine 5mg will be injected intravenously.

CONTACTS AND LOCATIONS:
Overall Officials: Sira Bang, MD PhD, Principal Investigator — Inje University Seoul Paik Hospital, Seoul, Korea
Locations (1):
- Inje University Seoul Paik Hospital, Seoul, Korea, Seoul, Jung-Gu,, South Korea